CLINICAL TRIAL: NCT01436565
Title: A Phase 1b Dose-escalation Study of the Safety and Pharmacokinetics of SAR245408 Administered in Combination With SAR256212 in Patients With Solid Tumor Cancers
Brief Title: A Study of Investigational SAR256212 in Combination With SAR245408 in Patients With Solid Tumor Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11721; U1111-1121-4146 (Other: UTN)
Record Dates: First submitted 2011-09-07; First posted 2011-09-19 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Solid Tumor Cancers
MeSH Terms: interventions — seribantumab; XL147

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dose escalation and expansion (Experimental): SAR245408 taken every day in the morning: no eating 2 hours prior and 1 hour after dose; SAR256212 will be given weekly by IV infusion over 1 hour, right after the SAR245408 oral dose
  Interventions: Drug: MM-121 (SAR256212); Drug: SAR245408

INTERVENTIONS:
Drug: MM-121 (SAR256212) — Pharmaceutical form:solution
  Route of administration: Intravenous
Drug: SAR245408 — Pharmaceutical form:tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

* To determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of SAR245408 administered in combination with SAR256212 in adult patients with locally advanced or metastatic solid tumors.

Secondary Objectives:

* To characterize the global safety profile of SAR245408 in combination with SAR256212
* To evaluate the pharmacokinetic (PK) profile of SAR245408 and SAR256212 used in combination
* To evaluate the objective response rate (ORR) and tumor volume change (for expansion cohort only)
* To determine the immunogenicity of SAR256212 as administered with SAR245408

DETAILED DESCRIPTION:
There is a 28 day screening period followed by 28 day cycles (21 day cycle for the every three week dosing regimen, if used) . Patients will continue to receive SAR245408/SAR256212 as long as there is clinical benefit or until a study withdrawal criterion is met. The last posttreatment visit will be 60 days after the last dose or until IMP-related toxicities have resolved or are deemed irreversible, whichever is later.

ELIGIBILITY:
Inclusion criteria:

* Metastatic or locally advanced nonhematological cancer, for which no alternative therapy is available
* Written informed consent
* For dose expansion only:

  * Patient's tumor harbors activating mutations in phosphoinositide-3-kinase, catalytic, alpha polypeptide (PIK3CA)
  * Tissue from archived sample
* Measurable and evaluable disease

Exclusion criteria:

* Patient less than 18 years old
* ECOG (Eastern Cooperative Oncology Group) performance status >2
* Any serious active disease or comorbid condition, which, in the opinion of the Investigator, could interfere with the safety of the patient or the ability of the patient to comply with the study, or with the interpretation of the results
* Poor bone marrow reserve as defined by absolute neutrophils count <1.5 x 109/L or platelets <100 x 109/L
* Poor organ function as defined by 1 of the following:

  * Total bilirubin >1.5 x ULN (upper limit of normal)
  * AST (aspartate aminotransferase) and/or ALT (alanine aminotransferase) >2.5 x ULN
  * Serum creatinine >1.5 x ULN and/or creatinine clearance <60 mL/min
  * PT/ (INR) (prothrombin time) (International Normalized Ratio) and/or partial thromboplastin time (PTT) test results ≥1.3 ULN
* Pregnant or breast-feeding women
* No use of effective birth control methods, when applicable
* No resolution of all specific toxicities (excluding alopecia) related to any prior anticancer therapy to Grade ≤1 according to the NCI common terminology criteria for adverse events (CTCAE) v.4.0
* Any of the following within 6 months prior to enrollment: myocardial infarction, severe/unstable angina, or coronary/peripheral artery bypass graft surgery, clinically symptomatic and uncontrolled cardiovascular disease, or clinically significant cardiac arrhythmias (Grade 3/4)
* Baseline corrected QT interval (QTc) >460 ms.
* NYHA Class III (New York Heart Association) or IV congestive heart failure or LVEF (left ventricular ejection fraction) < the lower limit of normal (LLN) for institution
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (including cytomegalovirus, Epstein-Barr virus, toxoplasmosis, and hepatitis B and C, positive for the human immunodeficiency virus (HIV), hypertension, or uncontrolled diabetes.
* Previous treatment with a selective PI3K inhibitor (phosphoinositide-3-kinase, catalytic, alpha polypeptide), mTOR (mechanistic target of rapamycin) inhibitor, or AKT inhibitor (v-akt murine thymoma viral oncogene homolog 1)
* Known hypersensitivity to the investigational medicinal product(s) or to its excipients, or patient who has had hypersensitivity reactions to fully human monoclonal antibodies
* Cytotoxic chemotherapy (including investigational cytotoxic agents) or biologic agents (antibodies, immune modulators, cytokines) within 4 weeks, or nitrosoureas or mitomycin C within 6 weeks, before the first dose of study treatment
* Prior radiation therapy within 2 weeks before the first dose of study treatment
* Prior major surgery from which the patient has not recovered or stabilized
* Any other investigational therapy within 4 weeks prior to the first dose of study treatment
* Brain tumor or brain metastasis are considered eligible if the patient has not received radiation therapy for brain metastasis within 2 weeks of enrollment and has been on a stable dose of steroids for 2 or more weeks
* Ongoing anticoagulation with therapeutic doses of warfarin (low-dose warfarin ≤1 mg/day is permitted).
* HBA1C (hemoglobin A1c) >7 or any patient requiring medication for glycemic control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 2 months to 12 months

SECONDARY OUTCOMES:
Peak and trough levels of SAR256212 and SAR245408 | 1 month to 6 months
Pharmacodynamic change in ErbB3 protein and mRNA levels as well as components of the PI3K pathway will be measured | 1 month to 6 months
Number of participants with adverse events | 1 month to 2 years
overall response rate | 2 months to 2 years
Number of patients who develop anti-MM-121 antibodies | 1 month to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840001, Boston, Massachusetts
  - Investigational Site Number 840101, Brookline, Massachusetts
  - Investigational Site Number 840002, Nashville, Tennessee